CLINICAL TRIAL: NCT05640154
Title: Health Promoting Lifestyle Program for Geriatric Patients' at Risk for Stroke
Brief Title: HPL Program for Geriatric Patients' at Risk for Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, TA Shoulkamy, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HPLgeriatric
Record Dates: First submitted 2022-11-03; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Health-Related Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational program (Experimental): aged patients 60 years and more, able to communicate, diagnosed with hypertension, diabetes mellitus and cardiac diseases. they will receive the nursing educational program which will be implemented in small groups from (5-7) in outpatient clinics. It includes nutrition, exercise, control hypertension , engage in weight control measures, smoking cessation, stress management, breathing exercise, appropriate treatment of diseases, control of diabetes, control of cholesterol in blood and routine follow up).also they will receive health-promoting lifestyle that includes (spiritual growth, interpersonal relations, nutrition, physical activity, health responsibility and stress management).
  Interventions: Behavioral: educational program
- control group (No Intervention): aged patients 60 years and more, able to communicate, diagnosed with hypertension, diabetes mellitus and cardiac diseases. the will not receive educational program and life style promotion.

INTERVENTIONS:
Behavioral: educational program — The nursing educational program will be implemented in small groups from (5-7) in outpatient clinics. It includes nutrition, exercise, control hypertension , engage in weight control measures, smoking cessation, stress management, breathing exercise, appropriate treatment of diseases, control of diabetes, control of cholesterol in blood and routine follow up).
  Arms: Educational program

SUMMARY:
Stroke is a highest reason of illness and death all over world. In 2017, stroke was the second greatest recurrent reason of mortality, after ischemic cardiac illness, and produced 6.2 million mortality all over world. The load of stroke does not only lie in the great mortality but the great morbidity also results in up to 50% of survivors being chronically disabled. Thus stroke is a disease of huge public health importance with economic and social consequences.

DETAILED DESCRIPTION:
Patients with stroke with uncontrolled glucose levels have higher mortality and poor post stroke outcomes. Controlling diabetes and other associated risk factors are effective ways to prevent initial strokes as well as stroke recurrence. Diabetes increases ischemic stroke incidence in all age groups, individuals with diabetes are more likely to suffer from hypertension, myocardial infarction and high cholesterol than individuals without diabetes have been linked to a greater risk of stroke. Smoking is a major cause of cardiovascular disease and causes one of every four deaths from cardiovascular disease. Smoking can raise triglycerides (a type of fat in your blood), Lower "good" cholesterol (high-density lipoprotein), Make blood sticky and more likely to clot, which can block blood flow to the heart and brain, Damage cells that line the blood vessels, Increase the buildup of plaque (fat, cholesterol, calcium, and other substances) in blood vessels and cause thickening and narrowing of blood vessels.The idea of lifestyle includes a broad variety of subjects, containing substantial life, spiritual life and other issues. Physical activity, smoking, alcohol consumption, nutrition and other aspects to measure lifestyle used by Chinese scientists. Health promoting lifestyle (HPL) is defined as "a multi-dimensional pattern of self-initiated actions and perceptions that serve to maintain or enhance the level of wellness, self-actualization, and fulfillment of the individual". It assesses a personal well-being activity that involves physical activity, dieting, spiritual growth, interpersonal relationships, health responsibility, and stress management, and would lead to enhaning wellbeing condition

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years and more
* Diagnosed with hypertension, diabetes mellitus and cardiac diseases.
* Able to communicate with health team, free from mental problems, and agreed to participate in the study were included.

Exclusion Criteria:

* unable to communicate with health team.
* free from mental problems.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-12-16 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
the effect of implementing nursing educational program on Health Promoting Lifestyle for geriatric patients' at risk for stroke. | 3 months
  by using tool II: It is a well-established instrument to assess personal lifestyle behaviors that promote health. It is composed of a 52-items questionnaire that is answered according to a 4-point Likert-type scale, with (Never (N) = 1, Sometimes (S) = 2, Often (O) = 3, Routinely (R) = 4). The total scale is 52-items and composed of six subscales to measure dimensions of health-promoting lifestyle that includes (spiritual growth, interpersonal relations, nutrition, physical activity, health responsibility and stress management). The total score will be adjusted from 0 to 100 and can classify the result to good lifestyle behavior if the percent score 60% and more and bad lifestyle behavior if less than 60%.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Asyut, Egypt